CLINICAL TRIAL: NCT06653361
Title: Ultra-Widefield Fluorescein Angiography-Based Targeted Retinal Photocoagulation Versus Conventional Panretinal Photocoagulation in the Preservation of Visual Function and Regression of Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hayatabad Medical Complex (Other Government)
Collaborators: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Yousaf Jamal Mahsood, Associate Professor, Hayatabad Medical Complex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 306/DME/KMC
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Proliferative Diabetic Retinopathy - High Risk
Keywords: Diabetic retinopathy; Laser photocoagulation; Fluorescein angiography
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRP (Experimental): Targeted Retinal Photocoagulation
  Interventions: Procedure: Green laser
- PRP (Active Comparator): Panretinal Photocoagulation
  Interventions: Procedure: Green laser

INTERVENTIONS:
Procedure: Green laser — Green Laser

SUMMARY:
Proliferative diabetic retinopathy is a vision-threatening disease that can lead to irreversible visual loss. The treatment options for proliferative diabetic retinopathy are anti-VEGF injection and retinal photocoagulation. The study aims to compare ultra-widefield fluorescein angiography-based targeted retinal photocoagulation and panretinal photocoagulation in the treatment of proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* proliferative diabetic retinopathy (PDR) with neovascularization on the disc or elsewhere in the retina

Exclusion Criteria:

* Participants with a history of previous history of:
* retinal photocoagulation
* vitreoretinal surgery
* tractional retinal detachment
* epiretinal membrane
* vitreomacular traction
* glaucoma
* uveitis
* media opacities like cataract, corneal opacity, vitreous hemorrhage
* anti-VEGF injections in last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
BCVA | 2 months
  Best Corrected Visual Acuity
CMT | 2 months
  Central Macular Thickness
MD | 2 months
  Mean Deviation
VFI | 2 months
  Visual Filed Index

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided